CLINICAL TRIAL: NCT04409314
Title: Pilot Study of Hypoxia-Specific Imaging to Predict Outcomes of Chimeric Antigen Receptor T-Cell Therapy
Brief Title: Hypoxia-Specific Imaging to Predict Outcomes of Chimeric Antigen Receptor T-cell Therapy
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 20921; NCI-2020-03216 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Aggressive Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent Malignant Neoplasm; Recurrent Plasma Cell Myeloma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Refractory Aggressive Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Malignant Neoplasm; Refractory Plasma Cell Myeloma; Refractory Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Multiple Myeloma; Neoplasms | interventions — fluoroazomycin arabinoside; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnostic (18F-FAZA PET scan): Prior to CAR T-cell therapy, patients receive administration of 18F-FAZA IV. Patients will then undergo a vertex-thigh PET scan approximately 2 hours after injection of 18FFAZA lasting 30-45 minutes.
  Interventions: Drug: Fluorine F 18-fluoroazomycin Arabinoside; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Fluorine F 18-fluoroazomycin Arabinoside — Given IV
  Other Names: 18F-FAZA; 18F-Fluoroazomycin Arabinoside; FAZA F-18; Fluoroazomycin Arabinoside F-18
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This study evaluates whether tumors present in patients with cancer who are planned to get CAR T-cells have low amounts of oxygen (hypoxia). PET scans may be used to check the amounts of oxygen within areas of cancer with a special radioactive tracer called FAZA that specifically looks for areas of low oxygen. This study is being done to help researchers determine how the amount of oxygen within areas of cancer affect how well CAR T-cells kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the incidence of intratumoral hypoxia in patients with relapsed or refractory (R/R) malignancies before treatment with chimeric antigen receptor (CAR) T-cell therapy.

SECONDARY OBJECTIVE:

I. To evaluate the association between intratumoral hypoxia and clinical responses to CAR T-cell therapy.

EXPLORATORY OBJECTIVES:

I. To correlate intratumoral hypoxia with markers of CAR T-cell activity and toxicity.

2. To correlate pre-therapy fluorine F 18-fluoroazomycin arabinoside (18F-FAZA) uptake with pre-therapy 18Ffluorodeoxyglucose (FDG) positron emission tomography (PET) uptake (if available).

OUTLINE:

Prior to CAR T-cell therapy, patients receive 18F-FAZA intravenously (IV). Beginning 2 hours after injection, patients undergo a single PET scan. Patients are followed for up to 6 months after CAR T-cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of:

  * Aggressive lymphoma, including: Diffuse large B-cell lymphoma (DLBCL) (including transformed disease), high-grade B-cell lymphoma, or primary mediastinal B-cell lymphoma
  * Multiple myeloma (MM), with imaging within 6 months of enrollment demonstrating >= 1 plasmacytoma measuring >= 5 cm along any axis
  * Other malignancy with radiographically measurable disease
* R/R disease with planned receipt of CAR T-cell therapy at University of California, San Francisco (UCSF), either through an Food and Drug Administration-approved CAR construct or through a separate interventional clinical trial
* Ability to provide informed consent prior to study entry

Exclusion Criteria:

* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with participant's safety, provision of informed consent, or compliance with study procedures
* Pregnancy or active lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed or refractory malignancies who are planning to receive CAR T-cell therapy at University of California, San Francisco (UCSF)
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Proportion of fluorine F 18-fluoroazomycin arabinoside (18F-FAZA) positron emission tomography (PET) scans with positive hypoxic volume (HV) | After completion of one-time 18F-FAZA PET scan, 1 day
  Will calculate the uniformly minimum-variance unbiased estimator, p-value and 95% confidence interval (CI) for the response rates.

SECONDARY OUTCOMES:
Overall response (OR) | At 30, 90, and 180 days after chimeric antigen receptor (CAR) T-cell therapy, up to 6 months
  Will determine OR at any time point as attainment of either complete response (CR) or partial response (PR). Logistic regressions will be used to evaluate the association between OR and intratumoral hypoxia, where hypoxia is analyzed as a binary and a continuous covariate.

OTHER OUTCOMES:
Change in Mean Serum Ferritin levels | Up to 6 months after CAR T-cell therapy
  Will use descriptive statistical methods to present data, including frequencies/percentages for categorical variables and means, medians, standard deviations, and ranges for continuous variables. Will evaluate the effect of intratumoral hypoxia and other exploratory endpoints using chi-squared tests and logistic regressions for categorical variables and two-sample t-tests and linear regressions for continuous variables.
Change in Mean C-reactive protein (CRP) levels | Up to 6 months after CAR T-cell therapy
  Will use descriptive statistical methods to present data, including frequencies/percentages for categorical variables and means, medians, standard deviations, and ranges for continuous variables. Will evaluate the effect of intratumoral hypoxia and other exploratory endpoints using chi-squared tests and logistic regressions for categorical variables and two-sample t-tests and linear regressions for continuous variables.
Change in Mean Fibrinogen Levels | Up to 6 months after CAR T-cell therapy
  Will use descriptive statistical methods to present data, including frequencies/percentages for categorical variables and means, medians, standard deviations, and ranges for continuous variables. Will evaluate the effect of intratumoral hypoxia and other exploratory endpoints using chi-squared tests and logistic regressions for categorical variables and two-sample t-tests and linear regressions for continuous variables.
Change in Hepatic aminotransferase Levels | Up to 6 months after CAR T-cell therapy
  Will use descriptive statistical methods to present data, including frequencies/percentages for categorical variables and means, medians, standard deviations, and ranges for continuous variables. Will evaluate the effect of intratumoral hypoxia and other exploratory endpoints using chi-squared tests and logistic regressions for categorical variables and two-sample t-tests and linear regressions for continuous variables.
Incidence of cytokine release syndrome (CRS), neurotoxicity, or other adverse events (AEs) attributed to CAR T-cell therapy | Up to 6 months after CAR T-cell therapy
  Will use descriptive statistical methods to present data, including frequencies/percentages for categorical variables and means, medians, standard deviations, and ranges for continuous variables. Will evaluate the effect of intratumoral hypoxia and other exploratory endpoints using chi-squared tests and logistic regressions for categorical variables and two-sample t-tests and linear regressions for continuous variables.
Standardized uptake value maximum (SUVmax) calculations for tumor sites based on 18F-FAZA versus fludeoxyglucose F-18 (18F-FDG) uptake | Up to 6 months after CAR T-cell therapy
  Will use descriptive statistical methods to present data, including frequencies/percentages for categorical variables and means, medians, standard deviations, and ranges for continuous variables. Will evaluate the effect of intratumoral hypoxia and other exploratory endpoints using chi-squared tests and logistic regressions for categorical variables and two-sample t-tests and linear regressions for continuous variables.

CONTACTS AND LOCATIONS:
Overall Officials: C. Babis Andreadis, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee R, Wang V, Huang CY, Pandita D, Leonard MK, LaRue S, Ahmadi M, Kaplan L, Ai WZ, Fakhri B, Spinner M, Seshadri MR, Pampaloni MH, Andreadis CB. Hypoxia-specific imaging in patients with lymphoma undergoing CAR-T therapy. Eur J Nucl Med Mol Imaging. 2023 Sep;50(11):3349-3353. doi: 10.1007/s00259-023-06296-z. Epub 2023 Jun 10. PMID 37300573